CLINICAL TRIAL: NCT00296738
Title: Quantitative 123I-MIBG SPECT/CT Assessment of Cardiac Sympathetic Innervation
Brief Title: 123I-MIBG SPECT/CT for Assessment of Cardiac Sympathetic Innervation
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. Alex Frenkel, Rambam Medical Center
Other Study IDs: MIBGCTIL
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Cardiac Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: SPECT/CT — GE INFINIA HAWKEYE

SUMMARY:
Myocardial scintigraphy with 123I-MIBG allows for visual and semi-quantitative assessment of sympathetic cardiac innervation using the hear to mediastinum ratio (HMR). Impaired cardiac MIBG clearance may occur in patients with congestive heart failure (CHF). The purpose of present study was to develop and validate a quantitative index for the assessment of cardiac MIBG uptake kinetics using SPECT/CT for diagnosis of CHF

ELIGIBILITY:
Inclusion Criteria:

* age>40

Exclusion Criteria:

* none

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients refered for neuroendocrine diseases
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The impact of the imaging modality on patient management | 2 years

SECONDARY OUTCOMES:
The impact on patient management | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Rispler, MD PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel